CLINICAL TRIAL: NCT01494116
Title: Factors Affecting Pediatric Isotonic Fluid Resuscitation Efficiency: Impact of Syringe Size
Brief Title: Pediatric Fast Fluid Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster Children's Hospital (Other)
Responsible Party: Principal Investigator, Melissa J Parker, MD, MSc, Assistant Professor, McMaster Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11-272
Record Dates: First submitted 2011-12-05; First posted 2011-12-16 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Fluid Resuscitation
Keywords: Pediatrics; Fluid; Bolus; Resuscitation; Shock
MeSH Terms: conditions — Shock | interventions — Saline Solution; Syringes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 10 mL syringe size (Experimental)
  Interventions: Other: 900 mL of 0.9% Normal Saline
- 20 mL syringe size (Experimental)
  Interventions: Other: 900 mL of 0.9% Normal Saline
- 30 mL syringe size (Experimental)
  Interventions: Other: 900 mL of 0.9% Normal Saline
- 60 mL syringe size (Experimental)
  Interventions: Other: 900 mL of 0.9% Normal Saline

INTERVENTIONS:
Other: 900 mL of 0.9% Normal Saline — The intervention consists of the administration of 900 mL of Normal Saline to the model using the "Disconnection- Reconnection" method of manual fluid resuscitation. All syringes (syringe size based on study arm) will be prepared by research staff following subject randomization. Each subject will take the prepared syringes, and sequentially administer them to the model by 1. Selecting and connecting a fluid-filled syringe to the catheter extension set to permit fluid administration 2. Manually administering the fluid to the model by depressing the syringe plunger 3. Disconnecting and discarding the empty syringe 4. Repeating steps 1-3 as fast as possible until all 900 mL has been administered.
  Other Names: BD 10 mL syringe with Luer-Lok Tip (Ref 309604); BD 20 mL syringe with Luer-Lok Tip (Ref 309661); BD 30 mL syringe with Luer-Lok Tip (Ref 309650); BD 60 mL syringe with Luer-Lok Tip (Ref 309653)

SUMMARY:
The purpose of this study is to determine the impact of syringe size on the amount of time it takes a health care provider to administer a known volume (900 mL) of resuscitation fluid to a non-clinical, toddler-sized, model. The investigators hypothesize that syringe size will impact fluid resuscitation time.

DETAILED DESCRIPTION:
The Surviving Sepsis Guideline for the resuscitation of pediatric septic shock indicates that up to 60 mL/kg of isotonic saline should be administered within the first 15 minutes of resuscitation. There are practical challenges to achieving these benchmarks. Syringes are often used to perform manual fluid resuscitation as they are generally available and health care providers are typically comfortable using them. Health care providers have been observed to have different preferences regarding the syringe size used to perform manual fluid resuscitation. Larger syringes e.g. 60 mL-size requires more force to depress the syringe plunger, due to a larger crosssectional area, but fewer syringes are needed to administer a given volume. Fewer syringes results in less time spent connecting and disconnecting syringes, which contributes to total fluid resuscitation time using this technique.

Consenting participants will be randomly assigned (by an independent Randomization Coordinator) to one of four syringe size groups (10 mL, 20 mL, 30 mL, 60 mL sizes). The allocation sequence is therefore concealed. After undergoing a standardization procedure, each participant will be instructed to administer 900 mL of 0.9% normal saline using pre-filled provided syringes by manual push as rapidly as possible using the disconnect-reconnect method. Participants will be advised to consider that they are in a situation where they are resuscitating a 15 kg child (represented by the model) in decompensated shock. Syringes for each 300 mL (20 mL/kg) aliquot will be colour-coded for identification purposes.

ELIGIBILITY:
Inclusion Criteria:

* Consenting health care staff and health care students capable of performing manual syringe bolus fluid administration

Exclusion Criteria:

* Non-English speaking individuals
* Any condition that would impact upon the individual's ability to perform manual fluid resuscitation e.g. limited hand strength or dexterity

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-10; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Total Intervention Time | From Date of Subject Randomization until Date Intervention Completed (Day 1)
  Subject is randomized and the intervention is performed the same day. Start Intervention Time (time zero): Subject begins administering the intervention; End Intervention Time: Subject has completed the intervention (900 mL of Saline has been administered); Total Intervention Time = End Intervention Time - Start Intervention Time. All testing is being video recorded. A blinded outcome assessor will review the video tapes and based upon clear, a priori defined, definitions will determine the Start Intervention Time and the End Intervention Time for each subject.

SECONDARY OUTCOMES:
Time to administer each of three sequential 300 mL fluid boluses | From Date of Subject Randomization until Date Intervention Completed (Day 1)
  Bolus 1 Time = Time at 300 mL administered MINUS Start Intervention Time; Bolus 2 Time = Time at 600 mL administered MINUS Time at 300 mL administered; Bolus 3 Time = Time at 900 mL administered (End Intervention Time) MINUS Time at 600 mL administered.
  Syringes are marked with coloured tape to facilitate identification according to Bolus number (Bolus 1 - Green; Bolus 2 - Yellow; Bolus 3 - Red).
Amount of normal saline actually administered to the model | From Date of Subject Randomization until Date Intervention Completed (Day 1)
  The normal saline administered to the model travels via conduit tubing in a dependent fashion to a graduated cylinder where it is collected for measurement upon completion of testing for each subject.
The proportion of subjects in each group that dislodge the IV catheter during testing. | From Date of Subject Randomization until Date Intervention Completed (Day 1)
  Any IV catheter dislodgement episodes will be recorded. The catheter used in this model is a 1.00 inch, 22-gauge, Insyte Autoguard IV catheter. The proximal end (hub) of the IV catheter is transfixed to the hand of the mannequin in typical clinical fashion, while the distal end is located within conduit tubing that leads to a 1 litre graduated cylinder. Connected to the hub of the IV catheter is a 7 inch long IV Catheter Extension Set.
Self-reported comfort of health care providers while performing the study intervention | From Date of Subject Randomization until Date Intervention Completed (Day 1)
  Based on responses to questionnaire that subjects are asked to complete following completion of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Melissa J Parker, MD, MSc, Principal Investigator — McMaster Children's Hospital
Locations (1):
- Hamilton Health Sciences, McMaster Children's Hospital, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Harvey G, Foster G, Manan A, Thabane L, Parker MJ. Factors affecting pediatric isotonic fluid resuscitation efficiency: a randomized controlled trial evaluating the impact of syringe size. BMC Emerg Med. 2013 Jul 24;13:14. doi: 10.1186/1471-227X-13-14. PMID 23883424